CLINICAL TRIAL: NCT02348892
Title: Evaluation Program of the Benefit of the Coordination of the Course of the Elderly Patient in Health Establishment - Pilot Study.
Acronym: PROCOPES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0343
Record Dates: First submitted 2015-01-16; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Elderly Patients in Complex Situations

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- With coordinator: Elderly patients, in complex situation, taken care by coordinator
  Interventions: Other: Coordinator
- Without coordinator: Elderly patients, in complex situation, taken care by the classic plan
  Interventions: Other: Classic plan

INTERVENTIONS:
Other: Coordinator — Patients in complex situation taken care by coordinator
  Groups: With coordinator
Other: Classic plan — Patients in complex situation taken care by classic plan
  Groups: Without coordinator

SUMMARY:
The large share of chronic diseases correlated with an aging population calls to develop necessary coordination between the hospital and non-hospital (professional of the city, home ...) to create new complementarities.

Since July 2013, the Nantes University Hospital experiences the establishment of a coordinator route patient in Gerontology. The evaluation program of the benefit of coordinating the course in elderly patients in health establishment (PROCOPES) must allow to prove the efficiency of the intervention of a coordinator route patient, following elderly patients in complex situations, both within the hospital and outside the hospital (home, nursing home,...). The objective of PROCOPES is to show the added value of an innovative position that can make the link between the hospital and the city on deemed complex situations.The pilot study results present a strong interest for health care settings, nursing home and in the world of research. It will also permit to have preliminary data for bigest studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient of 70 and more years old
* Patient living on Nantes
* Hospitalized in Nantes UH
* Patient whose the hospitalization is not relevant at the time of the request of trajectory case manager
* Patient whose the situation is complex (without solution at the time of the request)
* Patient (or legal representative) having given his assent of participation

Exclusion Criteria:

* Patient (or legal representative) refusing to participate in the protocol
* Patient whose follow-up is impossible (ex: programmed move, life expectation)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The eligible patients for the study will be the patients of 70 and more years old hospitalized in the Nantes UH in the acute care medical department internal medical departement medical urgency, rehabilitation unit, neurology, gastro-enterology of the CHU of Nantes and which are in complex medical and social situation, whoever is their motive for hospitalization.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Cost-utility analysis (CUA) | 6 months
  A differential cost-utility ratio will be used to compare both interventions. The evaluation of costs will take into account direct health care insurance cost, hospital costs and patient cost (according to the french health care insurance system). The evaluation of utility will be based on the evaluation of patient's quality of life, measured by EuroQol EQ-5D.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes UH, Nantes, France